CLINICAL TRIAL: NCT02858375
Title: Long-Term Assessment of Quality of Life and Effectiveness of Onabotulinumtoxina Injections in Provoked Vestibulodynia
Acronym: QUALVESTO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/175
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Vestibulodynia
Keywords: quality of life; botulinum toxin; provoked vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to assess and compare the pain in women suffering from provoked vestibulodynia, before treatment with botulinum injections, 3 months after treatment and 18 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Vestibulodynia rated B2 according to 2003 International Society for the Study of Vulvovaginal Disease (ISSVD) classification
* Patients previously treated no later than18 months ago for provoked vestibulodynia with botulinum toxin injections, in the University Hospital of Besançon.

Exclusion Criteria:

* Major psychologic disorders.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from provoked vestibulodynia, monitored in the Dermatology Department of the University Hospital of Besançon
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Long-term pain improvement after botulinum toxin injections | 18 months
  Assessment and comparison of pain using Visual Analogic Scale values before treatment,3 months after treatment and 18 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Pelletier, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France